CLINICAL TRIAL: NCT03581266
Title: Determination of Glucose Kinetics After Wheat and Rye Breads to Understand Their Physiological Effects
Brief Title: Glucose Kinetics After Wheat and Rye Breads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish University of Agricultural Sciences (Other)
Collaborators: Uppsala University (Other); CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Principal Investigator, Ali A Moazzami, Associate professor, PhD, Swedish University of Agricultural Sciences
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2014/290
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus, Type 2. Physiology of Glucose Kinetics
Keywords: Rye; Wheat; Rye factor; Glucose kinetics
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study was carried out using a crossover design with a three-week washout period. The participants stayed overnight at the facility and had one out of two types of breakfast in the morning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rye (Experimental): A breakfast consisting of whole slices of wholemeal rye bread containing 50 g of available carbohydrates. The breakfast additionally included 250 mL water and 50 g of cucumber.
  Interventions: Other: Rye/Wheat
- Wheat (Experimental): A breakfast consisting of whole slices of refined wheat bread containing 50 g of available carbohydrates. The breakfast additionally included 250 mL water and 50 g of cucumber.
  Interventions: Other: Rye/Wheat

INTERVENTIONS:
Other: Rye/Wheat — Mechanistic study of glucose kinetics after ingestion two kinds of bread

SUMMARY:
Certain functional properties of cereal products, e.g. their postprandial glucose and insulin responses, have been characterized as steps towards obtaining a greater understanding of their beneficial health effects. A low-glycemic index diet results in decreased postprandial insulin and glucose responses, which is thought to be beneficial for insulin and glucose metabolism.

In healthy subjects, it has been shown that rye breads (RBs) produce a lower postprandial insulin response compared with refined wheat breads (RWB) despite similar glucose responses. Juntunen et al. (2003) suggested that the difference in the structural characteristics between rye and wheat breads is a possible explanatory mechanism. However, the underlying mechanism of this discrepancy between insulin and glucose responses to rye bread, the so-called "rye factor" (RF), is still largely unknown. Faster starch digestibility and higher postprandial insulin responses for RWB compared with RBs may indicate faster intestinal glucose absorption and faster glucose disappearance respectively.

Therefore our hypothesis is that despite having similar glucose responses, RWB has faster turn over (kinetics) compared with RBs. The present study is aiming to apply an experimental set up which can comprehend the hypothetical differences in RWB and RBs kinetics.

DETAILED DESCRIPTION:
The human subjects after an overnight fasting 10-12 hours are coming to the clinic. On arrival, catheters are inserted into a forearm vein of each arm for blood sampling and isotope infusion, respectively. A primed followed by a constant-rate infusion of [6,6-2H2] glucose are administered. The enrichment of [6,6-2H2] glucose in the blood is then measured at different time points after the breakfast. The glucose kinetics can be calculated from this.

ELIGIBILITY:
Inclusion Criteria:

* Males 18-40 years with BMI 22-25.5 kg/m2

Exclusion Criteria:

* A family history of diabetes mellitus, regular use of nicotine, recurrent extensive exercise, regular intake of medication or food intolerances. The subjects had to be free from illnesses for one month prior to the study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only males were recruited
Enrollment: 10 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Investigate glucose kinetics after ingestion of wheat and rye breads | Completed and published study within 3 years after end of sample collection
  Glucose kinetics are investigated after ingestions of two different kinds of bread based breakfasts in order to see how the body responds to the different breads.

CONTACTS AND LOCATIONS:
Overall Officials: Ali A Moazzami, PhD, Principal Investigator — Swedish University of Agricultural Sciences

IPD SHARING:
Plan to Share IPD: Undecided